CLINICAL TRIAL: NCT02037542
Title: A Study of Lifestyle Intervention in Overweight or Obese Women With Early Stage Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Responsible Party: Principal Investigator, Michelle Gallas, Clinical Research Administrator, Baptist Health South Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 072013
Record Dates: First submitted 2013-07-16; First posted 2014-01-16 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Weight
Keywords: BMI, Lipid profile
MeSH Terms: conditions — Body Weight | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diet and Exercise (Experimental): Prospective, observational, cohort study, with a proposed start date of May 2013 and proposed end date of June 2018. Our goal is to gather data on a total of 200 patients: 100 patients (study group) will be prospectively enrolled, while data on another 100 patients (control) will be accessed through retrospective data collection. Number of patients to be analyzed will depend on enrollment and patient compliance. We would like to enroll the proposed 100 patients in the first 1-3 years of the study (approximately 30 per year).
  Interventions: Behavioral: Diet and exercise

INTERVENTIONS:
Behavioral: Diet and exercise — Upon enrollment, the patient will be asked to meet with a dietitian to assess the individual patient's current diet and exercise routines. In the first session, the dietitian will provide individual counseling and together with the patient devise weight loss / exercise strategies that fit the patients' lifestyle. Following the initial assessment, patients will embark on a weekly program, with weekly meetings lasting 30min - 1h. Patients will be asked to record meal portions weekly in a Food Log (Appendix B), according to the established goal. At each meeting, the dietitian will review the Food Log with the patient and evaluate progress.

SUMMARY:
The purpose of this study is to test the hypothesis that an intervention of lifestyle modification will positively impact women with breast cancer who are overweight and/or obese. To that end, our primary endpoint is to examine the effects of a practical lifestyle intervention that can be implemented by overweight or obese women (BMI greater or equal to 25) with early stage breast cancer (I-III) on outcomes such as body weight and change in BMI over the course of the study.

DETAILED DESCRIPTION:
* Primary endpoint: To examine the effects of a practical lifestyle intervention that can be implemented by overweight or obese women (BMI greater or equal to 25) with early stage breast cancer (I-III) on outcomes such as body weight and change in BMI over the course of the study.
* Secondary endpoint: To assess the impact of such intervention on lipid profiles and hemoglobin A1C. The study group will be compared with a historical control group of patients with early stage breast cancer who are obese or overweight who were not given the intervention
* Secondary endpoint: To examine whether an active intervention program will lead into longstanding lifestyle modification in breast cancer patients with a BMI greater or equal to 25.

ELIGIBILITY:
Inclusion Criteria:

* DCIS
* Women with stage 0 - III breast cancer (histologic type ductal or lobular)
* BMI >=25
* Patients must have completed all chemotherapy
* Patients may be on hormonal therapy or radiation therapy
* Age >= 18 years old to 89 Years old
* Patient must be medically stable and without significant impairments that would preclude following the proposed intervention regimen.
* Time of diagnosis: patients enrolled are within 1 month to 18 months post-diagnosis.

Exclusion Criteria:

* Metastatic breast cancer patients and patients with inoperable or active loco-regional disease.
* Patients following alternative/complementary diets or taking high dose antioxidant supplements.
* Patients with a physical/psychiatric impairment that would seriously impair their physical mobility.
* Patients who are currently suffering from severe nausea, anorexia or other diseases affecting health (e.g. arthritis and multiple sclerosis).
* Patients younger than 18 and older than 89 years.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Lifestyle intervention | One year
  To examine the effects of a practical lifestyle intervention that can be implemented by overweight or obese women (BMI greater or equal to 25) with early stage breast cancer (I-III) on outcomes such as body weight and change in BMI over the course of the study.

SECONDARY OUTCOMES:
Lipid Profiles, hemoglobin A1C | 1 year
  To assess the impact of such intervention on lipid profiles and hemoglobin A1C. The study group will be compared with a historical control group of patients with early stage breast cancer who are obese or overweight who were not given the intervention and to examine whether an active intervention program will lead into longstanding lifestyle modification in breast cancer patients with a BMI greater or equal to 25.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Amelia Rodrigues, MD, Principal Investigator — BHSF
Locations (1):
- South Miami Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dignam JJ, Wieand K, Johnson KA, Fisher B, Xu L, Mamounas EP. Obesity, tamoxifen use, and outcomes in women with estrogen receptor-positive early-stage breast cancer. J Natl Cancer Inst. 2003 Oct 1;95(19):1467-76. doi: 10.1093/jnci/djg060. PMID 14519753
- [Background] Christy SM, Mosher CE, Sloane R, Snyder DC, Lobach DF, Demark-Wahnefried W. Long-term dietary outcomes of the FRESH START intervention for breast and prostate cancer survivors. J Am Diet Assoc. 2011 Dec;111(12):1844-51. doi: 10.1016/j.jada.2011.09.013. PMID 22117660
- [Background] Demark-Wahnefried W, Morey MC, Sloane R, Snyder DC, Miller PE, Hartman TJ, Cohen HJ. Reach out to enhance wellness home-based diet-exercise intervention promotes reproducible and sustainable long-term improvements in health behaviors, body weight, and physical functioning in older, overweight/obese cancer survivors. J Clin Oncol. 2012 Jul 1;30(19):2354-61. doi: 10.1200/JCO.2011.40.0895. Epub 2012 May 21. PMID 22614994